CLINICAL TRIAL: NCT02056301
Title: A Comparison Trial Between Patient Controlled Intravenous Analgesia (PCA) and Epidural Analgesia for Pectus Excavatum Repair
Brief Title: A Comparison Trial Between PCA and Epidural Analgesia for Pectus Excavatum Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: New method of pain control pushed by surgeons.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Chris Glover, Pediatric Anesthesiologist, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H31096
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest | interventions — Hydromorphone; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Controlled Analgesia (Active Comparator): One group will have a patient controlled device connected to an intravenous patient controlled analgesia (IV PCA). This device runs a basal infusion of pain medicine (morphine) intravenously with additional allowable patient controlled doses every 10 minutes.
  Interventions: Drug: Morphine
- epidural Catheter (Active Comparator): The other group will have an epidural catheter inserted under sterile conditions in the thoracic epidural space after anesthesia has been induced. This will be connected to a patient controlled epidural analgesia (PCEA) device for postoperative pain control that works in a similar manner except the medication (a combination of local anesthetics and hydromorphone) will be administered in the thoracic epidural space.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — In keeping with standard practice at the TCH, the position of the thoracic epidural catheter tip will be confirmed by real time fluoroscopy and a single injection of 1 ml of omnipaque 180 mg/mL contrast. In keeping with current practice, a bolus of 0.2% ropivacaine 0.3 ml per kg (maximum dose 20 ml) will be administered in the epidural space to the patients in the TEA group at least 10 minutes prior to surgical incision.
  Arms: epidural Catheter
Drug: Morphine — This device runs a basal infusion of pain medicine (morphine) intravenously with additional allowable patient controlled doses every 10 minutes
  Arms: Patient Controlled Analgesia

SUMMARY:
The aim of this study is to compare the efficacy of epidural and IV analgesia in controlling pain in patients undergoing Nuss repair of pectus excavatum. The primary end point will be the mean pain score during postoperative days 0-4.

DETAILED DESCRIPTION:
Pectus excavatum is a cartilaginous deformity that is the most common congenital anterior chest wall defect in children [1]. Children with this disease process often complain of dyspnea, decreased exercise tolerance, and shortness of breath implying a restrictive pulmonary deficit [2]. Besides the reported physical limitations, patients can also exhibit manifestations of psychological disturbances (poor body image and depression). Surgical repair has been correlated with enhanced quality of life and improvement in body image[3] with recent studies showing improved pulmonary function and cardiac output [4, 5]. Surgery initially introduced by Sauerbruch involved rib cartilage resection and sternal osteotomy. This open procedure was further modified and became [6] known as the Ravitch procedure. This was the mainstay for repair for over 40 years until the introduction of minimally invasive surgery without rib resection by Nuss and colleagues in 1987 [7]. The Nuss repair involves placing an intrathoracic brace through small lateral chest wall incisions aided by thoracoscopy. Similar to bracing the teeth, the Nuss procedure avoids osteotomy or rib cartilage resection [8]. The Nuss procedure is the most common minimally invasive procedure in use today to correct this condition and is the current standard of surgical practice. Complications from Nuss repair can range anywhere from 7% to 25% [9] and can occur for as long as the bar is in place. Pain control remains a major issue in the perioperative period as patients may require weeks to months of oral narcotics before becoming pain-free after correction of the pectus. A prospective multicenter study reported peak pain scores of 8 on a 0-10 scale in the postoperative period and a mean score of 3 at discharge [4]. Postoperative pain after pectus repair has been managed with IV opioids administered by patient controlled analgesia (PCA) devices and by thoracic epidural infusions of combinations of local anesthetics and opioids. It is unclear from published data which method is superior and different tertiary care centers in the USA have a preference for different methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 8- 18 years 2) Patients undergoing minimally invasive pectus excavatum repair via Nuss procedure 3) American Society of Anesthesiology Status I-III

Exclusion Criteria:

* 1) Refusal of epidural catheter 2) Pregnancy 3) Bleeding History 4) Inability to understand how to use the PCA device 5) Medication interfering with blood coagulation 6) Patients allergic to local anesthetics 7) Patient refusal to participate in study 8) Developmental delay

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08; Primary Completion 2019-04-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Glover, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children't Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Controlled Analgesia | Epidural Catheter
Started | 33 | 29
Completed | 31 | 23
Not Completed | 2 | 6
Not completed — Protocol Violation | 1 | 2
Not completed — Surgical complications req. 2nd surgery | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Issues with epidural | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Controlled Analgesia | Epidural Catheter | Total
Number analyzed (Participants) | 31 | 23 | 54
Age, Continuous [Mean (Full Range); unit: years] — Age on day of surgery
  years | 15.7 [12.6 to 17.7] | 16.0 [12.9 to 17.8] | 15.8 [12.6 to 17.8]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 26 | 21 | 47
  Female | 3 | 1 | 4
  Unknown | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 23 | 54
ASA Status [Count of Participants; unit: Participants] — The ASA Physical Status Classification System assesses a patient's pre-anesthesia medical co-morbidities. The scale ranges from 1 to 6 with lower scores indicating a healthier patient. This is measured during the pre-operative assessment.
  Participants
    ASA I | 8 | 7 | 15
    ASA II | 20 | 15 | 35
    ASA III | 1 | 0 | 1
    ASA IV | 0 | 0 | 0
    ASA V | 0 | 0 | 0
    ASA VI | 0 | 0 | 0
    Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Scale Scores During Postoperative Days 0-4
Description: The aim of this study is to compare the efficacy of epidural and IV analgesia in controlling pain in patients undergoing Nuss repair of pectus excavatum. The primary end point will be the mean pain scores during postoperative days (POD) 0-4. Pain was measured using the verbal pain scale. The scale ranges from 0-10. A score of 0 means the patient is in no pain.
Time Frame: Postoperative days 0-4
Population: Pain scores could not be collected on each post-operative day because some subjects were discharged from the hospital quicker than others.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Controlled Analgesia | Epidural Catheter
Number analyzed (Participants) | 29 | 21
units on a scale
  Post-Operative Day 0: number analyzed (Participants) | 28 | 20
  Post-Operative Day 0 | 3.69 (1.98) | 2.28 (1.63)
  Post-Operative Day 1: number analyzed (Participants) | 28 | 19
  Post-Operative Day 1 | 2.77 (2.19) | 1.11 (1.18)
  Post-Operative Day 2 | 2.25 (1.65) | 2.14 (1.8)
  Post-Operative Day 3: number analyzed (Participants) | 21 | 21
  Post-Operative Day 3 | 2.69 (1.33) | 2.73 (1.85)
  Post-Operative Day 4: number analyzed (Participants) | 16 | 19
  Post-Operative Day 4 | 2.24 (1.52) | 2.14 (2.5)

2. Secondary Outcome: Total Morphine Equivalent Consumption During Postoperative Days 0-4
Description: This outcome measures total amount of morphine administered in mg/kg by post-operative day 0-4. This captures all standard of care opioids delivered via their assigned cohort route (Epidural vs. IV PCA). Opioids other than morphine that were administered for pain were multiplied by their equianalgesic conversion factor to calculate the IV Morphine equivalent.
Time Frame: Postoperative days 0-4
Population: Total Morphine Equivalent Consumption could not be collected on each post-operative day for every subject because some subjects were discharged from the hospital quicker than others.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Patient Controlled Analgesia | Epidural Catheter
Number analyzed (Participants) | 31 | 23
mg/kg
  Day 0 | 0.75 (0.34) | 0.14 (0.06)
  Day 1 | 0.90 (0.42) | 0.23 (0.12)
  Day 2 | 0.67 (0.33) | 0.61 (0.34)
  Day 3: number analyzed (Participants) | 29 | 23
  Day 3 | 0.57 (0.36) | 0.92 (0.23)
  Day 4: number analyzed (Participants) | 19 | 21
  Day 4 | 0.39 (0.32) | 0.45 (0.34)

3. Secondary Outcome: Rescue Morphine Equivalent Administration During Postoperative Days 0-4
Description: This outcome measures the amount of rescue morphine administered due to breakthrough pain in mg/kg by post-operative day 0-4. This captures additional opioids that were administered by a nurse through an IV. Opioids other than morphine that were administered for pain were multiplied by their equianalgesic conversion factor to calculate the IV Morphine equivalent.
Time Frame: Postoperative days 0-4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Patient Controlled Analgesia | Epidural Catheter
Number analyzed (Participants) | 31 | 23
mg/kg
  Day 0 | 1.26 (0.89) | 0.57 (0.73)
  Day 1 | 0.23 (0.67) | 0.26 (0.69)
  Day 2 | 0.13 (0.50) | 0.70 (1.15)
  Day 3: number analyzed (Participants) | 29 | 23
  Day 3 | 0.07 (0.26) | 0.39 (0.94)
  Day 4: number analyzed (Participants) | 19 | 21
  Day 4 | 0.05 (0.23) | 0.10 (0.44)

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events until hospital discharge, up to postoperative day 4.
Arm/Group | Patient Controlled Analgesia | Epidural Catheter
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/29
Other Adverse Events (participants affected / at risk) | 3/33 | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Controlled Analgesia (N=33) | Epidural Catheter (N=29)
Surgical Complications (Surgical and medical procedures) | 1 (1) | 0 — Surgical complications requiring secondary surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Controlled Analgesia (N=33) | Epidural Catheter (N=29)
Epidural Related (Surgical and medical procedures) | 3 (3) | 3 (3) — Epidural Placement Failed or Epidural Dislodged and subject switched to IV PCA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02056301/Prot_SAP_000.pdf